CLINICAL TRIAL: NCT01923376
Title: Hepatic Encephalopathy: Lactulose or Polyethylene Glycol (H.E.L.P.)
Acronym: HELP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough staff to collect data
Sponsor: New York Presbyterian Brooklyn Methodist Hospital (Other)
Responsible Party: Principal Investigator, Smruti R Mohanty, MD, Chief of Gastroenterology, New York Presbyterian Brooklyn Methodist Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 401550
Record Dates: First submitted 2013-07-25; First posted 2013-08-15 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Hepatic Encephalopathy; HE; Cirrhosis; Altered Mental Status; AMS
Keywords: hepatic encephalopathy; hepatic coma; HE; PSE; lactulose; golytely; cirrhosis; Hepatic Insufficiency; Liver Cirrhosis; Fibrosis; Brain Damage, Chronic; Delirium; Encephalitis; Neurotoxicity Syndromes; Liver Failure; Liver Diseases; Digestive System Diseases; Brain Diseases, Metabolic; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Metabolic Diseases; Pathologic Processes; Confusion; Neurobehavioral Manifestations; Neurologic Manifestations; Signs and Symptoms; Delirium, Dementia, Amnestic, Cognitive Disorders; Mental Disorders; Central Nervous System Viral Diseases; Virus Diseases; Central Nervous System Infections; Poisoning; Substance-Related Disorders; Citric Acid
MeSH Terms: conditions — Hepatic Encephalopathy; Fibrosis; Hepatic Insufficiency; Liver Cirrhosis; Brain Damage, Chronic; Delirium; Encephalitis; Neurotoxicity Syndromes; Liver Failure; Liver Diseases; Digestive System Diseases; Brain Diseases, Metabolic; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Metabolic Diseases; Pathologic Processes; Confusion; Neurobehavioral Manifestations; Neurologic Manifestations; Signs and Symptoms; Neurocognitive Disorders; Mental Disorders; Central Nervous System Viral Diseases; Virus Diseases; Central Nervous System Infections; Poisoning; Substance-Related Disorders | interventions — Lactulose; polyethylene glycol 3350; Golytely

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactulose (Other): per standard of care
  Interventions: Drug: Lactulose
- polyethylene glycol 3350 (Golytely) (Active Comparator)
  Interventions: Drug: Polyethylene Glycol 3350

INTERVENTIONS:
Drug: Lactulose — If randomized to this group, subjects will receive 10 - 30 grams of lactulose per standard of care
  Other Names: Enulose, Duphalac, generlac, kristalose
  Arms: Lactulose
Drug: Polyethylene Glycol 3350 — If subject is randomized to this group, one time dose of one gallon polyethylene glycol 3350 will be given at the time of enrollment
  Other Names: Miralax; Golytely
  Arms: polyethylene glycol 3350 (Golytely)

SUMMARY:
The purpose of this study is to evaluate whether the use of polyethylene glycol is superior and more safe in treating hepatic encephalopathy compared to lactulose and also to determine if treatment with polyethylene glycol will reduce the duration of hospital stay.

DETAILED DESCRIPTION:
Hepatic encephalopathy is the occurrence altered level of consciousness as a result of cirrhosis and liver failure. Main treatment goal for hepatic encephalopathy is to eliminate the precipitating factor and to decrease circulating ammonia level. Current standard for treating HE is treatment with Lactulose. Lactulose are metabolized by colonic bacteria to byproducts which cause catharsis and reduces pH, thereby inhibiting ammonia absorption. However, there is limited evidence available to demonstrate the efficacy. Studies on animal model have suggested that polyethylene glycol 3350-electrolyte solution (GOLYTELY) is effective in clearing gut bacteria and reducing the ammoniagenesis in colon. Recently published study by Robert Rahimi, University of Texas Southwestern Medical Center found that polyethylene glycol is more effective in improving HE over the first 24 hours compared to lactulose and also may reduce duration of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 80
* Male and female of all races and ethnicities
* Cirrhosis of any cause
* Any grade of hepatic encephalopathy (1-4)
* Representatives have to be willing to comply with all protocol procedures and to understand, sign and date an informed consent document and authorize access to protected health information on the subject's behalf

Exclusion Criteria:

* Acute liver failure
* Prisoners
* Structural brain lesions (as indicated by CT and confirmed by neurological exam)
* Other causes of altered mental status
* Previous use of rifaximin or neomycin within last 7 days
* Pregnancy
* Serum Na <125 MEq/liter
* Receiving more than 1 dose (30 cc) of lactulose prior to enrollment
* Uncontrolled infection with hemodynamic instability requiring vasopressors.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Improvement of cognition | 24 hours from the time of enrollment
  Subjects will be evaluated every 24hr from the time of enrollment to assess for improvement of cognition until back to baseline and/or grade 0 based on HESA scare

SECONDARY OUTCOMES:
Duration of hospital stay | From time of admission to time of discharge an approximate length of seven days
  To determine if treatment with polyethylene glycol compared to lactulose will reduce the duration of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Smruti R Mohanty, MD, Principal Investigator — New York Presbyterian Brooklyn Methodist Hospital
Locations (1):
- New York Methodist Hospital, Brooklyn, New York, United States